CLINICAL TRIAL: NCT01512264
Title: Post-Stroke Aphasia and rTMS Treatment Study (PART)
Brief Title: Post-Stroke Aphasia and Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment Study
Acronym: PART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Jerzy P Szaflarski, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01HD068488 (NIH)
Record Dates: First submitted 2012-01-10; First posted 2012-01-19 (Estimated); Results first posted 2019-08-16 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Aphasia; Stroke
Keywords: Aphasia; Stroke; functional Magnetic resonance imaging; fMRI; Language recovery after stroke; constraint induced aphasia therapy; CIAT; Repetitive transcranial magnetic stimulation; rTMS
MeSH Terms: conditions — Aphasia; Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- rTMS (Experimental): 3 weeks of nerTMS
  Interventions: Device: Magstim SuperRapid
- 1 week of Sham Treatment + 2 weeks of nerTMS (Sham Comparator): 1 week of Sham Treatment + 2 weeks of nerTMS
  Interventions: Device: Magstim SuperRapid
- 2 weeks of Sham Treatment +1 week of nerTMS (Sham Comparator): 2 weeks of Sham Treatment +1 week of nerTMS
  Interventions: Device: Magstim SuperRapid
- Control Group (Placebo Comparator): 3 weeks of Sham Treatment
  Interventions: Device: Magstim SuperRapid

INTERVENTIONS:
Device: Magstim SuperRapid — This design will allow systematic evaluation of the efficacy of nerTMS and its most optimal dose for language recovery.
  Other Names: Repetitive Transcranial Magnetic Stimulation, rTMS

SUMMARY:
In this study the investigators will examine the efficacy of navigated excitatory repetitive transcranial magnetic stimulation (nerTMS) for the treatment of post stroke aphasia. The investigators expect that this new types of rehabilitation (nerTMS) will help patients with aphasia return to their lives as they were prior to the stroke.

DETAILED DESCRIPTION:
Aphasia after stroke is associated with high mortality, significant motor impairment, and severe limitations in social participation. During the past decade, therapies administered by stroke teams have made great strides to limit the motor impairments caused by stroke. Unfortunately, progress in aphasia rehabilitation has not experienced the same rapid advancement. This proposal is based on preliminary evidence from our recently completed pilot study which showed that navigated excitatory repetitive transcranial magnetic stimulation (nerTMS) targeted to residual activity in the affected hemisphere has a significant beneficial effect on post-stroke aphasia recovery.1 The main aim of this study is to conduct a double-blind, sham-controlled, dose-response nerTMS treatment trial in subjects with chronic aphasia. By conducting this comparative trial, we will provide clinical (qualitative and quantitative) and imaging evidence that nerTMS improves language function after stroke when compared to standard treatment (ST). The findings will have implications for patients with post-stroke aphasia in that once the study is completed and the results are available, rehabilitation specialists may be able to change their practice pattern by offering an additional tool to aid patients in recovering their language skills with improved participation in society and enhanced quality of life.

To fill the gap in our therapeutic arsenal for aphasia, we propose a study with the following specific aims: (1) to determine the comparative efficacy and optimal dosing of nerTMS on aphasia recovery using a randomized, double-blind, sham-controlled study design. Subjects (15/group) will be randomly assigned to 4 treatment groups: (a) 3 weeks of nerTMS, (b) 1 week of ST + 2 weeks of nerTMS, (c) 2 weeks of ST +1 week of nerTMS, or (d) 3 weeks of ST (control group). This design will allow systematic evaluation of the efficacy of nerTMS and will determine its most optimal dose for language recovery. Short- and long-term outcomes will be evaluated with aphasia testing (AT) and fMRI; (2) to use fMRI to assess changes in language lateralization in response to nerTMS. We will examine the relationship between the degree of pre-nerTMS language lateralization (fMRI) with the post-nerTMS language outcomes (AT) and determine whether fMRI language lateralization can predict AT performance following nerTMS targeted to the left middle cerebral artery (LMCA) stroke areas.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* LMCA stroke as indicated by the presence of aphasia and MRI lesion in the LMCA distribution
* Moderate aphasia (Token Test score between 40th and 90th percentile)
* Fluency in English
* Provision of written informed consent by the patient and/or the next of kin

Exclusion Criteria:

* Age less than 18 years
* Underlying degenerative or metabolic disorder or supervening medical illness
* Severe depression or other psychiatric disorder
* Positive pregnancy test in women of childbearing age
* Any contraindication to MRI/fMRI at 3T (i.e., intracranial metal implants, claustrophobia)
* Any contraindication to nerTMS (e.g., seizures or epilepsy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-01; Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy P Szaflarski, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Started | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 6
Not Completed | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group | Total
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 3 | 7 | 22
  >=65 years | 1 | 1 | 4 | 0 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 1 | 8
  Male | 4 | 6 | 4 | 6 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 3 | 9
  White | 5 | 5 | 4 | 4 | 18
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 6 | 7 | 27
  India | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Aphasia Testing as Evaluated by the Boston Naming Test (BNT) - Baseline
Description: 60-item test of visual confrontation naming for aphasia. In the BNT, subjects are shown line drawings of common objects one at a time and asked to name them orally. Scoring counts the number of spontaneously produced correct responses, the number of cues given, and the number of responses after phonemic cuing and after semantic cuing. The scale for scoring is 0-60 with 0 being no spontaneous correct answers and 60 being all correct answers.
Time Frame: Baseline: 1 week before the first nerTMS treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
units on a scale | 33.43 (17.67) | 18.29 (18.94) | 28.57 (24.21) | 41.00 (13.56)

2. Primary Outcome: Aphasia Testing as Evaluated by the Boston Naming Test (BNT) - Immediate Follow-Up
Description: as for outcome 1
Time Frame: within 1 week post treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
units on a scale | 42.43 (18.32) | 24.86 (22.23) | 30.86 (24.65) | 48.83 (10.26)
Statistical Analysis 1: Comparison: rTMS; paired t- test between time point 1 and time point 4 for the rTMS group and BNT test was calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -1.58; Test type: Other; p = 0.006, t-test, 2 sided
Statistical Analysis 2: Comparison: 1 Week of Sham Treatment + 2 Weeks of nerTMS; paired t- test between time point 1 and time point 4 for the1 week of Sham Treatment + 2 weeks of nerTMS group and BNT test was calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -1.27; Test type: Other; p = 0.015, t-test, 2 sided
Statistical Analysis 3: Comparison: 2 Weeks of Sham Treatment +1 Week of nerTMS; paired t- test between time point 1 and time point 4 for the 2 weeks of Sham Treatment + 1 week of nerTMS group and BNT test was calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -0.54; Test type: Other; p = 0.203, t-test, 2 sided
Statistical Analysis 4: Comparison: Control Group; paired t- test between time point 1 and time point 4 for the control group and BNT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -1.63; Test type: Other; p = 0.010, t-test, 2 sided

3. Primary Outcome: Aphasia Testing as Evaluated by the Boston Naming Test (BNT) - Long Term Follow-up
Description: as for outcome 1
Time Frame: 3 months post treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
units on a scale | 38.50 (20.44) | 15.67 (17.69) | 25.17 (24.69) | 47.60 (9.56)
Statistical Analysis 1: Comparison: rTMS; paired t- test between time point 1 and time point 5 for the rTMS group and BNT test was calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -0.54; Test type: Other; p = 0.410, t-test, 2 sided
Statistical Analysis 2: Comparison: 1 Week of Sham Treatment + 2 Weeks of nerTMS; paired t- test between time point 1 and time point 5 for 1 week of Sham Treatment + 2 weeks of nerTMS group and BNT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = 0.57; Test type: Other; p = 0.618, t-test, 2 sided
Statistical Analysis 3: Comparison: 2 Weeks of Sham Treatment +1 Week of nerTMS; paired t- test between time point 1 and time point 5 for 2 weeks of Sham Treatment + 1 week of nerTMS group and BNT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = 1.31; Test type: Other; p = 1.000, t-test, 2 sided
Statistical Analysis 4: Comparison: Control Group; paired t- test between time point 1 and time point 5 for the control group and BNT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = 4.35; Test type: Other; p = 0.019, t-test, 2 sided

4. Primary Outcome: Aphasia Testing as Evaluated by the Semantic Fluency Test (SFT) - Baseline
Description: The Semantic Fluency Test is used to assess verbal ability. It is a psychological test where participants produce as many words as possible in a given category for a specified time period. In the SFT participants were given 3 categories (i.e. "Animals", "Fruits") and asked to produce as many words in that category as they can in 60 seconds. Scoring of the test included the sum of the number of spontaneous words that were generated in each category. This measure does not have a theoretical maximum; however, the more words generated indicates higher verbal ability which can indicate changes related to aphasia.
Time Frame: 1 week before the first nerTMS treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: words generated
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
words generated | 16.29 (13.01) | 8.00 (7.66) | 9.57 (9.03) | 25.50 (8.92)

5. Primary Outcome: Aphasia Testing as Evaluated by the Semantic Fluency Test (SFT) - Immediate Follow-up
Description: as for outcome 4
Time Frame: within 1 week post treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
units on a scale | 18.86 (13.43) | 8.86 (8.76) | 11.14 (10.11) | 29.17 (9.58)
Statistical Analysis 1: Comparison: rTMS; paired t- test between time point 1 and time point 4 for the rTMS group and SFT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -0.69; Test type: Other; p = 0.118, t-test, 2 sided
Statistical Analysis 2: Comparison: 1 Week of Sham Treatment + 2 Weeks of nerTMS; paired t- test between time point 1 and time point 4 for the 1 week of Sham Treatment + 2 weeks of nerTMS group and SFT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -0.28; Test type: Other; p = 0.482, t-test, 2 sided
Statistical Analysis 3: Comparison: 2 Weeks of Sham Treatment +1 Week of nerTMS; paired t- test between time point 1 and time point 4 for the 2 weeks of Sham Treatment +1 week of nerTMS group and SFT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -0.37; Test type: Other; p = 0.368, t-test, 2 sided
Statistical Analysis 4: Comparison: Control Group; paired t- test between time point 1 and time point 4 for the control group and SFT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -0.70; Test type: Other; p = 0.147, t-test, 2 sided

6. Primary Outcome: Aphasia Testing as Evaluated by the Semantic Fluency Test (SFT) - Long Term Follow-up
Description: as for outcome 4
Time Frame: 3 months post treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: words generated
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
words generated | 19.00 (12.86) | 7.50 (8.87) | 9.83 (9.39) | 30.40 (5.32)
Statistical Analysis 1: Comparison: rTMS; paired t- test between time point 1 and time point 5 for the rTMS group and SFT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -0.54; Test type: Other; p = 0.410, t-test, 2 sided
Statistical Analysis 2: Comparison: 1 Week of Sham Treatment + 2 Weeks of nerTMS; paired t- test between time point 1 and time point 5 for the 1 week of Sham Treatment + 2 weeks of nerTMS group and SFT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = 0.25; Test type: Other; p = 0.695, t-test, 2 sided
Statistical Analysis 3: Comparison: 2 Weeks of Sham Treatment +1 Week of nerTMS; paired t- test between time point 1 and time point 5 for the 2 weeks of Sham Treatment +1 week of nerTMS group and SFT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -0.25; Test type: Other; p = 0.175, t-test, 2 sided
Statistical Analysis 4: Comparison: Control Group; paired t- test between time point 1 and time point 5 for the control group and SFT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -0.60; Test type: Other; p = 0.518, t-test, 2 sided

7. Primary Outcome: Aphasia Testing as Evaluated by the Controlled Word Association Test (COWAT) - Baseline
Description: The Controlled Word Association Test is also a verbal fluency test. In this test participants produce as many words as possible given a specific letter for a specified time period. In the COWAT participants were given 3 Letters (i.e. "C", "F", "L") and asked to produce as many words that begin with that letter (excluding proper nouns) as they can in 60 seconds. Scoring of the test included the sum of the number of spontaneous words that were generated in each category. This measure does not have a theoretical maximum; however, the more words generated indicates higher verbal ability which can indicate changes related to aphasia.
Time Frame: 1 week before the first nerTMS treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: words generated
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
words generated | 9.29 (8.14) | 4.43 (6.24) | 4.86 (3.98) | 9.33 (5.68)

8. Primary Outcome: Aphasia Testing as Evaluated by the Controlled Word Association Test (COWAT) - Immediate Follow-up
Description: as for outcome 7
Time Frame: within 1 week post treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: words generated
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
words generated | 12.43 (10.13) | 5.43 (5.53) | 5.00 (5.35) | 10.17 (5.56)
Statistical Analysis 1: Comparison: rTMS; paired t- test between time point 1 and time point 4 for the rTMS group and COWAT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -0.71; Test type: Other; p = 0.109, t-test, 2 sided
Statistical Analysis 2: Comparison: 1 Week of Sham Treatment + 2 Weeks of nerTMS; paired t- test between time point 1 and time point 4 for the 1 week of Sham Treatment + 2 weeks of nerTMS group and COWAT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -0.28; Test type: Other; p = 0.485, t-test, 2 sided
Statistical Analysis 3: Comparison: 2 Weeks of Sham Treatment +1 Week of nerTMS; paired t- test between time point 1 and time point 4 for the 2 weeks of Sham Treatment +1 week of nerTMS group and COWAT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -0.07; Test type: Other; p = 0.864, t-test, 2 sided
Statistical Analysis 4: Comparison: Control Group; paired t- test between time point 1 and time point 4 for the control group and COWAT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -0.43; Test type: Other; p = 0.341, t-test, 2 sided

9. Primary Outcome: Aphasia Testing as Evaluated by the Controlled Word Association Test (COWAT) - Long Term Follow-up
Description: as for outcome 7
Time Frame: 3 months post treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: words generated
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
words generated | 9.67 (8.38) | 3.33 (4.18) | 4.67 (5.47) | 12.60 (5.50)
Statistical Analysis 1: Comparison: rTMS; paired t- test between time point 1 and time point 5 for the rTMS group and COWAT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -0.12; Test type: Other; p = 0.899, t-test, 2 sided
Statistical Analysis 2: Comparison: 1 Week of Sham Treatment + 2 Weeks of nerTMS; paired t- test between time point 1 and time point 5 for the 1 week of Sham Treatment + 2 weeks of nerTMS group and COWAT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = 0.19; Test type: Other; p = 0.519, t-test, 2 sided
Statistical Analysis 3: Comparison: 2 Weeks of Sham Treatment +1 Week of nerTMS; paired t- test between time point 1 and time point 5 for the 2 weeks of Sham Treatment +1 week of nerTMS group and COWAT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -0.09; Test type: Other; p = 1.000, t-test, 2 sided
Statistical Analysis 4: Comparison: Control Group; paired t- test between time point 1 and time point 5 for the control group and COWAT test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -0.84; Test type: Other; p = 0.140, t-test, 2 sided

10. Primary Outcome: Western Aphasia Battery (WAB) - Baseline
Description: WAB assesses linguistic skills most frequently affected by aphasia, plus key nonlinguistic skills, and provides differential diagnosis information. Adaptable to various administration settings from hospital room to clinic, it provides a baseline level of performance to measure change over time.The scoring provides two main totals, in addition to the subscale scores. These are the Aphasia Quotient (AQ) score and Cortical Quotient (CQ) score. AQ can essentially be thought of as a measure of language ability, whilst CQ is a more general measure of intellectual ability and includes all the subscales. Administration of the Western Aphasia Battery (WAB) yields a total score termed the Aphasia Quotient (AQ), which is said to reflect the severity of the spoken language deficit in aphasia. This score is a weighted composite of performance on 10 separate WAB subtests. Scores rate severity as follows: 0-25 is very severe, 26-50 is severe, 51-75 is moderate, and 76-above is mild.
Time Frame: Baseline: 1 week before the first nerTMS treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
units on a scale | 64.214 (33.201) | 54.883 (28.649) | 54.380 (27.405) | 81.740 (13.639)

11. Primary Outcome: Western Aphasia Battery (WAB) - Immediate Follow-Up
Description: as for outcome 10
Time Frame: within 1 week post treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
units on a scale | 63.500 (36.559) | 51.520 (27.751) | 57.460 (28.076) | 77.700 (12.895)
Statistical Analysis 1: Comparison: rTMS; paired t- test between time point 1 and time point 4 for the rTMS group and WAB test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = 0.24; Test type: Other; p = 0.520, t-test, 2 sided
Statistical Analysis 2: Comparison: 1 Week of Sham Treatment + 2 Weeks of nerTMS; paired t- test between time point 1 and time point 4 for the 1 week of Sham Treatment + 2 weeks of nerTMS group and WAB test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = 0.97; Test type: Other; p = 0.800, t-test, 2 sided
Statistical Analysis 3: Comparison: 2 Weeks of Sham Treatment +1 Week of nerTMS; paired t- test between time point 1 and time point 4 for the 2 weeks of Sham Treatment +1 week of nerTMS group and WAB test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -0.68; Test type: Other; p = 0.148, t-test, 2 sided
Statistical Analysis 4: Comparison: Control Group; paired t- test between time point 1 and time point 4 for the control group and WAB test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = 0.67; Test type: Other; p = 0.787, t-test, 2 sided

12. Primary Outcome: Western Aphasia Battery (WAB) - Long-Term Follow-Up
Description: as for outcome 10
Time Frame: 3 months post treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
units on a scale | 72.417 (31.692) | 50.560 (27.219) | 61.960 (31.587) | 84.425 (12.807)
Statistical Analysis 1: Comparison: rTMS; paired t- test between time point 1 and time point 5 for the rTMS group and WAB test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -3.12; Test type: Other; p = 0.239, t-test, 2 sided
Statistical Analysis 2: Comparison: 1 Week of Sham Treatment + 2 Weeks of nerTMS; paired t- test between time point 1 and time point 5 for the 1 week of Sham Treatment + 2 weeks of nerTMS group and WAB test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = 2.71; Test type: Other; p = 0.212, t-test, 2 sided
Statistical Analysis 3: Comparison: 2 Weeks of Sham Treatment +1 Week of nerTMS; paired t- test between time point 1 and time point 5 for the 2 weeks of Sham Treatment +1 week of nerTMS group and WAB test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -3.10; Test type: Other; p = 0.120, t-test, 2 sided
Statistical Analysis 4: Comparison: Control Group; paired t- test between time point 1 and time point 5 for the control group and WAB test were calculated. Cohen's d was calculated to determine the power of the test. The Cohen's d calculated for this test = -1.14; Test type: Other; p = 0.263, t-test, 2 sided

13. Secondary Outcome: Change in Language Laterilazation as Indicated by Neuroimaging Correlates: Frontal Laterality Index (LI) Scores - Baseline
Description: Laterality index (LI) is a measure of language lateralization to a hemisphere - it ranges from "-1" (or -100%) indicating left-hemispheric lateralization to "1" (or 100%) indicating right-hemispheric lateralization. A change from the baseline visit to the post-treatment visit is a neuroimaging (fMRI) outcome measure in this study. Change in LI does not indicate improvement or worsening but rather shift in lateralization of the language function representation in the brain that may be correlated with change in linguistic testing (e.g., WAB).
Time Frame: Baseline: 1 week before the first nerTMS treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: Index score
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
Index score | 0.30 (0.40) | 0.22 (0.20) | -0.19 (0.30) | 0.13 (0.42)

14. Secondary Outcome: Change in Language Lateralization as Indicated by Neuroimaging Correlates: Frontal Laterality Index (LI) Scores - Immediate Follow-up
Description: as for outcome 13
Time Frame: within 1 week post treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: index score
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
index score | 0.02 (0.40) | 0.09 (0.46) | -0.09 (0.55) | -0.01 (0.39)

15. Secondary Outcome: Change in Language Lateralization as Indicated by Neuroimaging Correlates: Frontal Laterality Index (LI) Scores - Long-term Follow Up
Description: as for outcome 13
Time Frame: 3 months post treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: index score
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
index score | 0.20 (0.41) | 0.20 (0.36) | 0.01 (0.69) | 0.20 (0.40)

16. Secondary Outcome: Change in Language Lateralization as Indicated by Neuroimaging Correlates: Frontal-Parietal Laterality Index (LI) Scores - Baseline
Description: as for outcome 13
Time Frame: Baseline: 1 week before the first nerTMS treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: index score
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
index score | 0.14 (0.21) | 0.15 (0.26) | -0.19 (0.22) | 0.10 (0.34)

17. Secondary Outcome: Change in Language Lateralization as Indicated by Neuroimaging Correlates: Frontal-Parietal Laterality Index (LI) Scores - Immediate Follow Up
Description: as for outcome 13
Time Frame: within 1 week post treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: index score
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
index score | 0.10 (0.31) | 0.06 (0.47) | -0.03 (0.46) | -0.03 (0.18)

18. Secondary Outcome: Change in Language Lateralization as Indicated by Neuroimaging Correlates: Frontal-Parietal Laterality Index (LI) Scores - Long-term Follow Up
Description: as for outcome 13
Time Frame: 3 months post treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: index score
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
index score | 0.21 (0.20) | -0.11 (0.14) | -0.02 (0.29) | 0.23 (0.23)

19. Secondary Outcome: Change in Language Lateralization as Indicated by Neuroimaging Correlates: Cerebellum Laterality Index (LI) Scores - Baseline
Description: as for outcome 13
Time Frame: Baseline: 1 week before the first nerTMS treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: index score
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
index score | -0.24 (0.23) | -0.05 (0.47) | -0.09 (0.33) | -0.23 (0.11)

20. Secondary Outcome: Change in Language Lateralization as Indicated by Neuroimaging Correlates: Cerebellum Laterality Index (LI) Scores - Immediate Follow Up
Description: as for outcome 13
Time Frame: within 1 week post treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: index score
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
index score | 0.06 (0.26) | -0.22 (0.35) | 0.01 (0.39) | -0.33 (0.42)

21. Secondary Outcome: Change in Language Lateralization as Indicated by Neuroimaging Correlates: Cerebellum Laterality Index (LI) Scores - Long-term Follow Up
Description: as for outcome 13
Time Frame: 3 months post treatment
Population: 1 participant from control group was unable to be analyzed due to loss of follow up.
Measure: Mean (Standard Deviation); unit: index score
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
Number analyzed (Participants) | 7 | 7 | 7 | 6
index score | -0.08 (0.35) | 0.02 (0.21) | 0.08 (0.20) | -0.28 (0.21)

ADVERSE EVENTS:
Time Frame: From baseline through 48 months
Description: 1 participant from control group was unable to be analyzed due to loss of follow up.
Arm/Group | rTMS | 1 Week of Sham Treatment + 2 Weeks of nerTMS | 2 Weeks of Sham Treatment +1 Week of nerTMS | Control Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT01512264/Prot_SAP_000.pdf